CLINICAL TRIAL: NCT03628664
Title: Preoperative CT Assisted Planning for Primary Total Knee Arthroplasty
Acronym: CT planning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Saeed Younis, Clinical investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 44556677
Record Dates: First submitted 2018-07-25; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT planned total knee arthroplasty (Active Comparator): Surgeon will follow the CT plan
  Interventions: Radiation: CT scan
- Non CT planned total knee arthroplasty (No Intervention): Surgeon will not follow the CT plan

INTERVENTIONS:
Radiation: CT scan — Assessment of the actual posterior condylar angle using the CT scan
  Arms: CT planned total knee arthroplasty

SUMMARY:
Total knee arthroplasty is one of the most common management methods of knee osteoarthritis. Patellar complications are one of the important causes of revision total knee arthroplasty. Proper placement of the components in the best rotational and axial alignment would achieve better patellar tracking and the best functional outcomes. Preoperative CT scan can add information regarding the coronal and rotational alignment of the prosthesis components.

DETAILED DESCRIPTION:
Total knee arthroplasty is the gold standard treatment for advanced knee osteoarthritis. In spite of the great advance in the prosthesis design, surgical techniques and rehabilitation programs, only 85% (75% to 92%) of patients with total knee arthroplasty are satisfied with their operations and 30% develops patellofemoral complications.

Femoral and tibial components malrotation is a crucial cause of postoperative knee pain, patellar instability, and may lead to revision. In measured resection technique the surgical epicondylar axis (SEA) is the center of rotation of the knee and the femoral component must be parallel to this axis. The surgical epicondylar axis is difficult to be determined intraoperative by palpation.

Commonly, surgeons routinely set the femoral posterior condyle resection at three degrees fixed from the posterior condylar line (PCL) because the PCL was found to be three degrees internally rotated from the (SEA).

The posterior condylar angle on a three-dimensional structure reconstruction of the CT scans in osteoarthritic knees has also been shown as 3.3° ± 1.5°, However, another study documented the posterior condylar angle (PCA) in osteoarthritic knees as 1.6° ± 1.9°. Also there is a two to three degree difference between the surgical epicondylar axis and the anatomical epicondylar axis. Therefore, a routine bone resection of three degrees from the PCL is not universal for all cases and may create malrotation of the femur.

CT scan can provide an adequate template with good but not excellent inter and intra observer reliability for exact determination of the surgical epicondylar axis and femoral component rotation.

2. AIM/ OBJECTIVES

1. What is the mean of distal femoral rotation in Egyptian population?
2. What is the effect of osteoarthritis on femoral rotation?
3. How much is the accuracy of CT scan in detecting anatomical landmarks to choose the intraoperative femoral component rotation (correlation between radiological and intraoperative findings?
4. Is the relation between the anatomical epicondylar axis (AEA) in comparison to surgical epicondylar axis (SEA) a fixed ratio?
5. What is the relation between thde femoral component malrotation and the coronal alignment and flexion gap balance?
6. Can CT scan add a simple planning tool for accurate placement of femoral component and the reproducibility of the preoperative plan in surgery?

ELIGIBILITY:
Inclusion Criteria:

* Advanced knee osteoarthritis in which total knee arthroplasty is indicated

Exclusion Criteria:

* Revision total knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Knee Society score (KSS) | one year
Western Ontario and McMaster university osteoarthritis index (WOMAC) score | One year

SECONDARY OUTCOMES:
Patient satisfaction: Knee Society score(KSS) subscale | one year
  Knee Society score(KSS) subscale satisfaction
Patellofemoral functional score | one year
  Barlett patellofemoral score
Revision rate | one year
  Number of patients undergoing revision knee arthroplasty surgery
Knee range of motion | one year
  Knee range of motion (flexion and extension)in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saeed Younis, Dr., Principal Investigator — Ain Shams University; Radwan Gamal Abdel Hamid, Dr., Study Director — Ain Shams University; Mohamed Awad, Dr., Study Director — Ain Shams University; Wael Samir Osman, professor, Study Chair — Ain Shams University; Tarek Mohammed Samy, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams Univrsity, Cairo, Egypt